CLINICAL TRIAL: NCT02216877
Title: Magnesium Supplementation for Hypomagnesemia in Chronic Kidney Disease - A Dose-Finding Trial
Brief Title: Magnesium Supplementation for Hypomagnesemia in Chronic Kidney Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Iain Bressendorff, Medical Doctor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MgCKDRos
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease; Hypomagnesemia
Keywords: Chronic Kidney Disease; Hypomagnesemia
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Magnesium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Oral placebo twice daily for 8 weeks. 12 subjects.
  Interventions: Drug: Placebo
- Mablet 360 mg once daily (Experimental): Oral Mablet 360 mg once daily and oral placebo once daily for 8 weeks. 12 subjects.
  Interventions: Drug: Mablet 360 mg; Drug: Placebo
- Mablet 360 mg twice daily (Experimental): Oral Mablet 360 mg twice daily for 8 weeks. 12 subjects.
  Interventions: Drug: Mablet 360 mg

INTERVENTIONS:
Drug: Mablet 360 mg
  Other Names: Magnesium hydroxide
  Arms: Mablet 360 mg once daily; Mablet 360 mg twice daily
Drug: Placebo
  Arms: Mablet 360 mg once daily; Placebo

SUMMARY:
Randomized placebo-controlled interventional trial to investigate the effect of oral magnesium supplementation on intracellular magnesium in subjects with chronic kidney disease. We hypothesize that oral magnesium supplementation will increase intracellular magnesium in subjects with chronic kidney disease as well as increase serum magnesium.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is associated with increase cardiovascular morbidity and mortality independent of traditional cardiovascular risk factors due to increased vascular calcification. Epidemiological and experimental data suggest that hypermagnesemia and magnesium supplementation reduce vascular calcification in chronic kidney disease by increasing calcium/phosphate solubility in serum, by inhibiting calcium influx into vascular smooth muscle cells (VSMC), by inhibiting intracellular pro-calcification enzymes in VSMC and by increasing activity of intracellular anti-calcification enzymes in VSMC. A trial to investigate the effect of oral magnesium supplementation on vascular calcification in subjects with CKD is currently being planned, but prior to initiating such a trial it is necessary to determine the dose of oral magnesium needed to increase intracellular magnesium and serum magnesium.

ELIGIBILITY:
Inclusion Criteria:

* Estimated Glomerular filtration rate (eGFR) < 60 mL/min.
* Serum magnesium < 0.82 mmol/L.
* Written informed consent.

Exclusion Criteria:

* Hemodialysis.
* Peritoneal dialysis.
* Kidney transplant recipient.
* Parathyroid hormone > 600 pg/L.
* Pregnancy.
* Comorbidity that makes study participation and completion impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Intracellular magnesium | 8 weeks
  Intracellular magnesium measured by energy dispersive x-ray analysis (www.exatest.com).

SECONDARY OUTCOMES:
Total serum magnesium | 8 weeks
Ionized serum magnesium | 8 weeks

OTHER OUTCOMES:
Markers of CKD-MBD (Chronic Kidney Disease - Mineral and Bone Disorder) | 8 weeks
  Serum calcium, phosphate, parathyroid hormone (PTH), fibroblast growth factor 23 (FGF-23), 25-(OH)-hydroxy vitamin D, 1,25-(OH)-dihydroxy vitamin D as well as urine calcium and phosphate.

CONTACTS AND LOCATIONS:
Overall Officials: Iain B Bressendorff, MD, Principal Investigator — Department of Medicine, Division of Nephrology, Roskilde County Hospital
Locations (1):
- Department of Medicine, Division of Nephrology, Roskilde County Hospital, Roskilde, Denmark